CLINICAL TRIAL: NCT03170128
Title: Functional Outcomes After Radial Head Fractures Treated Non-operatively
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-03464
Record Dates: First submitted 2017-05-26; First posted 2017-05-30 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Radial Head Fracture
MeSH Terms: conditions — Radial Head and Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient Physical Therapy (Active Comparator)
  Interventions: Procedure: Outpatient physical therapy in addition to standard follow-up visits
- Home Exercises (Active Comparator)
  Interventions: Behavioral: Home exercises in addition to standard follow-up visits

INTERVENTIONS:
Procedure: Outpatient physical therapy in addition to standard follow-up visits — Patients in Group 1 will be given a prescription for outpatient physical therapy.
  Arms: Outpatient Physical Therapy
Behavioral: Home exercises in addition to standard follow-up visits — Patients in Group 2 will be carefully instructed on home exercises for range of motion and strengthening of their affected elbow. All therapy regimens will be prescribed at initial presentation, as is the current practice. All other care will be identical for patients in both groups. This
  Arms: Home Exercises

SUMMARY:
The purpose of this study is to investigate the effects of physical therapy as part of the non-operative treatment of radial head fractures.There is currently no data to support the use of physical therapy in the non-operative treatment of radial head fractures. Likewise, there is no data that shows that physical therapy is harmful to patients being treated non-operatively for radial head fractures. Investigators believe that prescribing physical therapy for patients with non-displaced radial head fractures treated non-operatively is unnecessary, and that that it would be equally efficacious to teach patients simple stretching exercises that they could perform by themselves. Subjects will be randomized into 2 groups: Group 1 - Patients will be prescribed physical therapy within the first month following fracture; Group 2 - Patients will be given simple stretching exercises to perform at home and will not be given a prescription for physical therapy. Patients who agree to participate in this study and sign the informed consent will be randomly assigned to one of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals to be approached for participation in this study will include all adult (age > 18 years old) patients who are receiving or seeking medical care in the outpatient setting.

Exclusion Criteria:

* Patients who are initially determined to need surgical fixation of a radial head fracture will not be included in this study. There are no additional exclusion criteria.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-08-03 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Successful fracture union | 3 Months
  Demonstrated through x-rays

SECONDARY OUTCOMES:
Functional outcome score | 3 Months
  functional survey scores will demonstrate that physical therapy does not impact patient outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egol, MD, Principal Investigator — NYU Hospital for Joint Diseases
Locations (1):
- New York University School of Medicine, New York, New York, United States